CLINICAL TRIAL: NCT06339333
Title: Evaluation of ACT Now GAIN Later: a Psychologist Guided Self Help Video Parenting Programme Based on Principles of Acceptance and Commitment Therapy (ACT)
Brief Title: Evaluation of ACT Now GAIN Later
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University College Dublin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: RRECB0523EC
Record Dates: First submitted 2024-02-29; First posted 2024-04-01 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Psychological Flexibility; Child Behavior; Relationship, Parent Child; Well-Being, Psychological; Self-efficacy
MeSH Terms: conditions — Child Behavior; Psychological Well-Being | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: This quantitative study will be a two arm randomised control trial with an intervention group and waitlist group.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACT Now GAIN Later (Experimental): This group will receive a 7-week psychologist guided parenting intervention.
  Interventions: Behavioral: ACT Now GAIN Later
- Waitlist Group (Active Comparator): This group will receive pre and post measures but will not receive an intervention until after the final measures have been administered.
  Interventions: Other: Control Group

INTERVENTIONS:
Behavioral: ACT Now GAIN Later — ACT Now GAIN Later is a Psychologist Guided Self Help Parenting Programme. This has been developed by HSE Senior psychologist,. Dr. Michelle Howard to help parents manage challenging behaviors in their children. Parents of children who are referred to HSE Psychology Services with behavioural difficulties are invited to participate in this 7 week programme.
  Arms: ACT Now GAIN Later
Other: Control Group — Waitlist Group
  Arms: Waitlist Group

SUMMARY:
The goal of this Randomised Control Trial is to evaluate a Psychologist Guided Self Help Video Parenting Programme based on principles of Acceptance and Commitment Therapy (ACT)

The main questions it aims to answer are:

Primary Objectives

1. Is ACT Now GAIN Later: a Psychologist Guided Self Help Video Parenting Programme based on principles of ACT effective in increasing parental psychological flexibility (measured by Psy-Flex, tool which measures psychological flexibility)? Please find attached.
2. Is ACT Now GAIN Later: a Psychologist Guided Self Help Video Parenting Programme based on principles of ACT effective in decreasing child challenging behaviour (measured by the Eyberg Child Behavior Inventory)? Please find attached.

Secondary Objectives

1. Is ACT Now GAIN Later: an ACT based Parenting Programme, effective in improving parent-child relationships (measured by the Child-Parent Relationship Scale)? Please find attached.
2. Does ACT Now GAIN Later increase parental well-being as measured by (Depression Anxiety Stress Scale, Parenting Stress Index and Goal Based Outcome Tool)? Please find attached.
3. Does ACT Now GAIN Later increase parental self-efficacy (TOPSE and Parental Sense of Competence scale)? Please find attached.

Participants will complete a 7 week psychologist guided parenting intervention. Researchers will compare waitlist groups to see if there are differences in psychological flexibility, child behaviour, parent-child relationships, parental well-being or parental self-efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Parents of children from the ages of 3-12 will be included in this study.
* Parents of children with challenging behavior.

Exclusion Criteria:

* Parents of children outside of the age range 3-12 years old
* Parents of children who do not have challenging behavior

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2024-05-12 (Estimated); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Parental Psychological Flexibility | Pre and Post Intervention (week 1 and week 7 - end of the intervention). Also 3 and 6 months post intervention.
  Psy-Flex: The scale ranges from a minimum score of 6 to a maximum score of 30. Higher scores indicate higher levels of psychological flexibility.
Child Behaviour | Pre and Post Intervention (week 1 and week 7 - end of the intervention). Also 3 and 6 months post intervention.
  Eyberg Child Behaviour Inventory: The scale ranges from 0 - 36. Higher scores indicate more problematic behaviours at greater frequency. Norms also exist for clinical cut off's.

SECONDARY OUTCOMES:
Parent-Child Relationships | Pre and Post Intervention (week 1 and week 7 - end of the intervention). Also 3 and 6 months post intervention.
  Child-Parent Relationship Scale: There are two sub scales; closeness and conflict. On the closeness sub scale, higher scores indicate better/ more positive parent-child relationships. On the conflict sub scale, lower scores indicate less conflict and higher scores indicate more conflict in the relationship.
Parental Well-Being | Pre and Post Intervention (week 1 and week 7 - end of the intervention). Also 3 and 6 months post intervention.
  Depression Anxiety Stress Scale: Scale range is 0 - 42. Higher scores indicate more distress. Subscales for anxiety, depression and stress.
Parental Self-Efficacy | Pre and Post Intervention (week 1 and week 7 - end of the intervention). Also 3 and 6 months post intervention.
  Parental Sense of Competence Scale: Lower scores indicate lower parental sense of competence and high scores indicate high parental sense of competence.
Parental Self-Efficacy | Pre and Post Intervention (week 1 and week 7 - end of the intervention). Also 3 and 6 months post intervention.
  Parenting Stress Index: Scores range from 18-90. Lower scores indicate lower levels of parenting stress.

CONTACTS AND LOCATIONS:
Locations (1):
- Longford Primary Care Centre, Longford, Ireland

IPD SHARING:
Plan to Share IPD: No